CLINICAL TRIAL: NCT03617874
Title: PC4PrEP: Integrating Pre-Exposure Prophylaxis (PrEP) Into Primary Care
Brief Title: PC4PrEP: Integrating PrEP Into Primary Care
Acronym: PC4PrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: HIV Center for Clinical & Behavioral Studies at Columbia University (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015-5847; R01MH107297 (NIH)
Record Dates: First submitted 2018-04-19; First posted 2018-08-07 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Human Immunodeficiency Virus Transmission
Keywords: Pre-exposure prophylaxis; Human Immunodeficiency Virus; PrEP; Risk for HIV acquisition; PrEP candidacy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PC4PrEP- Intervention Clinics (Active Comparator): Intervention clinics will receive the PC4PrEP intervention. The intervention includes Montefiore PrEP policy awareness, provider and patient education, pre-screening to identify PrEP eligible patients, and identifying high risk individuals in the community and providing referral and linkage to primary care.
  Interventions: Other: PC4PrEP- Intervention Clinics
- Standard of Care Clinics (Placebo Comparator): These clinics will not receive the PC4PrEP intervention but will continue with their standard of care model.
  Interventions: Other: Standard of Care Clinics

INTERVENTIONS:
Other: PC4PrEP- Intervention Clinics — PC4PrEP is a comprehensive, multi-level, structural and sustainable intervention designed to address barriers at system, provider, and user levels to increase PrEP uptake.
  Arms: PC4PrEP- Intervention Clinics
Other: Standard of Care Clinics — The standard of care model is the model approved by the health system for their health care clinics.
  Arms: Standard of Care Clinics

SUMMARY:
Oral pre-exposure prophylaxis (PrEP) has been proven effective in reducing HIV infection in high-risk men who have sex with men, heterosexually active women and men, and injecting drug users. Despite its 2012 approval by the FDA and the development of Centers for Disease Control and Prevention (CDC) clinical guidelines, PrEP uptake has been limited. Significant impediments to PrEP implementation include: system barriers (lack of a medical "home" and of models for implementing PrEP); provider barriers (difficulty identifying those likely to benefit from PrEP, inexperience with PrEP, and concerns about adherence and risk compensation); and user barriers (lack of awareness of PrEP, inability to access providers comfortable with prescribing PrEP, and concerns about stigma and side effects). Cost is not a barrier in New York State, where PrEP is covered by many insurance plans, including Medicaid.

Primary Care for PrEP (PC4PrEP) is a structural, multilevel intervention that will integrate PrEP into primary care practices that care for underserved communities in the Bronx, NY, an epicenter of continuing HIV infection in the US. PC4PrEP will develop an organizational protocol for prescribing PrEP in primary care; identify high-risk individuals in primary care clinics and community HIV testing sites using a new PrEP Eligibility Tool; link them to primary care providers (PCPs) who can provide PrEP; and counsel potential users about PrEP both before they receive a prescription (to enhance receptivity), and after they initiate PrEP (to enhance adherence). In the course of this study, investigator(s) will (1) develop and pilot PC4PrEP; (2) implement and evaluate it in "real-world" settings (Federally Qualified Health Centers; FQHCs) on objective outcomes as well as provider and patient reports; and (3) present a new model, the PrEP Cascade that - as with the HIV Care Cascade for HIV+ populations - may be used to evaluate the impact of PrEP programs in the US and other countries. PC4PrEP is consistent with CDC and New York State Department of Health (NYSDOH) Guidelines and the Affordable Care Act in integrating PrEP into primary care practices and is responsive to recent 2014 NYSDOH recommendations which now position PrEP as a first-line intervention for MSM and transgender women who engage in ongoing anal sex without condoms, HIV- partners in sero-discordant relationships, and high-risk heterosexual women in high seroprevalence areas.There are two Specific Aims: (1) Finalize the PC4PrEP intervention and, in a clinic-randomized Phase 2 futility trial, assess whether it shows promise for increasing PrEP prescription rates in the Bronx, NY; and (2) Identify strengths and limitations of PC4PrEP in two ways: (a) through a mixed-methods process evaluation PrEP-eligible patients and PCPs, counselors and navigators; and (b) by identifying "fall-off" at each step of the PrEP Cascade.

DETAILED DESCRIPTION:
Primary Care for PrEP (PC4PrEP)

Although oral pre-exposure prophylaxis (PrEP) was approved by the FDA in 2012, and the CDC has developed interim clinical practice guidelines, uptake has been limited. The literature has identified system, provider, and user barriers to PrEP implementation. System barriers include lack of a medical home ("the purview paradox") and of organizational models for implementing PrEP. Provider barriers include difficulty identifying those likely to benefit from PrEP, inexperience with PrEP, and concerns about adherence and risk compensation. User barriers include lack of awareness of PrEP, inability to access providers who are comfortable prescribing it, and concerns about stigma and side effects. Cost is not a barrier in New York State (NYS), where PrEP is covered by many insurance plans, including Medicaid, and is provided to the uninsured. To date, real-world interventions to promote PrEP uptake for those at high risk of HIV acquisition have not been developed and formally evaluated. Implementation science research demonstration projects are urgently needed to determine the most effective strategies for integrating PrEP into primary care. The long term goal of PC4PrEP is to reduce the number of new HIV infections through developing a transferable model of PrEP delivery in primary care settings that are situated in high HIV incidence communities. The objective of this study is to develop, implement and evaluate Primary Care for PrEP (PC4PrEP), a new multilevel structural intervention that will address system, provider, and user barriers to PrEP uptake.

PC4PrEP has four components. It will: (1) designate a "home" for PrEP in primary care clinics; (2) train and support primary care providers (PCPs) to prescribe and manage PrEP, and create provider norms that promote the value of PrEP; (3) identify high-risk individuals in primary care clinics using a new PrEP Eligibility Tool developed by our team; and (4) identify high-risk out-of-care individuals (in collaboration with a community-based organization that conducts outreach and HIV testing in HIV-risk groups) and link them to PCPs who can provide PrEP. Investigator(s) will counsel potential users about PrEP both before they receive a prescription (to enhance receptivity), and after they initiate PrEP (to enhance adherence).

Investigator(s) will conduct a Phase 2 clinic-randomized futility trial of PC4PrEP in six Montefiore Medical Center Federally Qualified Health Centers (FQHCs) and a non-randomized Bronx Community Based Organization (CBO) to determine whether PC4PrEP shows promise for increasing the rate of new PrEP prescriptions, assess its effect on outcomes at each stage of our conceptualization of the "PrEP Cascade," and assess challenges to PrEP adoption.

The Specific Aims are:

1. Assess effects of PC4PrEP measured as the rate of new PrEP prescriptions per clinic per year;
2. Through a phased implementation of the four components of PC4PrEP, determine the incremental contribution of each component;
3. Evaluate the effects of PC4PrEP on measures of the "PrEP Cascade";
4. Assess challenges to PC4PrEP adoption through (1) in-depth interviews with PCPs and support staff about PC4PrEP; (2) in-depth interviews with selected patient-provider dyads to understand their communication about PrEP; (3) a nested longitudinal qualitative study of patients who initiate PrEP that will include exploration of risk compensation and self-reported adherence augmented by an objective measure of adherence, dried blood spot assays for tenofovir disphosphate.

Investigator(s) will develop, pilot, implement PC4PrEP; evaluate it in "real-world" settings (FQHCs) via objective outcomes as well as provider and patient reports. PC4PrEP will be developed by our multidisciplinary academic-community team from the Montefiore Medical Center, the Albert Einstein College of Medicine, the HIV Center for Clinical and Behavioral Studies at NYS Psychiatric Institute and Columbia University, and Bronx CBO. PC4PrEP is driven by Montefiore Medical Center policy (that PCPs promote PrEP); designed by those who will actually use it for seamless implementation, efficiency and sustainability; and uses existing staff in their current job titles and prevailing health care practices [e.g., electronic medical record (EMR) "best practice" alerts, screening tools, HIV counselors, continuing medical education].

ELIGIBILITY:
Inclusion Criteria:

* Patient at Montefiore Medical Center or Bronx Community Based Organization (CBO)
* Assessed to be eligible for PrEP by PCP
* Willing to provide dried blood spot (DBS) samples for antiretroviral anabolite testing
* Willing to provide access to medical records
* Willing to have interview audio-recorded
* No grossly evident cognitive impairment precluding consent and participation
* Speaks Spanish or English

Exclusion Criteria:

* Less than 18 years of age
* Not a patient at Montefiore Medical Center or Bronx Community Based Organization (CBO)
* Assessed to be ineligible for PrEP by PCP
* Unwilling to provide dried blood spot samples for ARV anabolite testing
* Unwilling to provide access to medical records
* Unwilling to have interview audio-recorded
* Unable to provide informed consent due to grossly evident cognitive impairment
* Does not speak Spanish or English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Rate of New PrEP Prescriptions | Up to12 months
  The primary outcome parameter of the trial is rate of new PrEP prescriptions/FQHC/year of observation. The primary quantitative outcome is the number of new PrEP prescriptions written in the past 12 months, determined when all PC4PrEP components have been implemented and in place for 12 months. The analysis will compare the rate of new PrEP prescriptions per clinic per year of observation in intervention and control clinics. We are not recruiting patients for this trial; outcomes are based on de-identified clinic data.

SECONDARY OUTCOMES:
Rate of Individuals at Risk for HIV Infection | Up to12 months
  The quantitative outcome is the number of HIV- individuals screened, and identified as potential PrEP candidates as assessed by the PrEP Eligibility Tool administered in the Intervention clinic. Outcomes are based on de-identified PrEP Eligibility Tool data.
Rate of Individuals Linked to Clinical Prevention | Up to 12 months
  The quantitative outcome is percentage of documented referrals or refusals by individuals being linked for clinical prevention.
Rate of Individuals Evaluated for PrEP | Up to 12 months
  PC4PrEP will educate, train, and mentor Primary Care Physicians to evaluate individuals for PrEP. The quantitative outcome is the percentage of individuals evaluated for PrEP, and PrEP eligibility as determined by providers.
Rate of PrEP Acceptance | Up to 12 months
  The quantitative outcome is the percentage of individuals who were interested in, accepted, initiated, or refused PrEP.
Rate of PrEP Adherence | Up to 12 months
  The quantitative outcome is the percentage of individuals adhering to PrEP and returning for medical follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie J. Bauman, PhD, Principal Investigator — Albert Einstein College of Medicine; Joanne Mantell, PhD, Principal Investigator — NYSPI HIV Center for Clinical & Behavioral Studies at Columbia University
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Interim guidance for clinicians considering the use of preexposure prophylaxis for the prevention of HIV infection in heterosexually active adults. MMWR Morb Mortal Wkly Rep. 2012 Aug 10;61(31):586-9. PMID 22874836
- [Background] Centers for Disease Control and Prevention (CDC). Update to Interim Guidance for Preexposure Prophylaxis (PrEP) for the Prevention of HIV Infection: PrEP for injecting drug users. MMWR Morb Mortal Wkly Rep. 2013 Jun 14;62(23):463-5. PMID 23760186
- [Background] Caceres CF, O'Reilly KR, Mayer KH, Baggaley R. PrEP implementation: moving from trials to policy and practice. J Int AIDS Soc. 2015 Jul 20;18(4 Suppl 3):20222. doi: 10.7448/IAS.18.4.20222. eCollection 2015. PMID 26198349
- [Background] Mantell JE, Sandfort TG, Hoffman S, Guidry JA, Masvawure TB, Cahill S. Knowledge and Attitudes about Pre-Exposure Prophylaxis (PrEP) among Sexually Active Men Who Have Sex with Men (MSM) Participating in New York City Gay Pride Events. LGBT Health. 2014 Mar 13;1(2):93-97. doi: 10.1089/lgbt.2013.0047. PMID 25346930
- [Background] Mimiaga MJ, Case P, Johnson CV, Safren SA, Mayer KH. Preexposure antiretroviral prophylaxis attitudes in high-risk Boston area men who report having sex with men: limited knowledge and experience but potential for increased utilization after education. J Acquir Immune Defic Syndr. 2009 Jan 1;50(1):77-83. doi: 10.1097/QAI.0b013e31818d5a27. PMID 19295337
- [Background] Arnold EA, Hazelton P, Lane T, Christopoulos KA, Galindo GR, Steward WT, Morin SF. A qualitative study of provider thoughts on implementing pre-exposure prophylaxis (PrEP) in clinical settings to prevent HIV infection. PLoS One. 2012;7(7):e40603. doi: 10.1371/journal.pone.0040603. Epub 2012 Jul 11. PMID 22792384
- [Background] Wheelock A, Eisingerich AB, Gomez GB, Gray E, Dybul MR, Piot P. Views of policymakers, healthcare workers and NGOs on HIV pre-exposure prophylaxis (PrEP): a multinational qualitative study. BMJ Open. 2012 Jul 2;2(4):e001234. doi: 10.1136/bmjopen-2012-001234. Print 2012. PMID 22761288
- [Background] Puro V, Palummieri A, De Carli G, Piselli P, Ippolito G. Attitude towards antiretroviral Pre-Exposure Prophylaxis (PrEP) prescription among HIV specialists. BMC Infect Dis. 2013 May 14;13:217. doi: 10.1186/1471-2334-13-217. PMID 23672424
- [Background] Krakower D, Mayer KH. Engaging healthcare providers to implement HIV pre-exposure prophylaxis. Curr Opin HIV AIDS. 2012 Nov;7(6):593-9. doi: 10.1097/COH.0b013e3283590446. PMID 23032736
- [Background] Krakower D, Ware N, Mitty JA, Maloney K, Mayer KH. HIV providers' perceived barriers and facilitators to implementing pre-exposure prophylaxis in care settings: a qualitative study. AIDS Behav. 2014 Sep;18(9):1712-21. doi: 10.1007/s10461-014-0839-3. PMID 24965676
- [Background] Hoffman S, Guidry JA, Collier KL, Mantell JE, Boccher-Lattimore D, Kaighobadi F, Sandfort TG. A Clinical Home for Preexposure Prophylaxis: Diverse Health Care Providers' Perspectives on the "Purview Paradox". J Int Assoc Provid AIDS Care. 2016 Jan-Feb;15(1):59-65. doi: 10.1177/2325957415600798. Epub 2015 Aug 20. PMID 26293904
- [Background] White JM, Mimiaga MJ, Krakower DS, Mayer KH. Evolution of Massachusetts physician attitudes, knowledge, and experience regarding the use of antiretrovirals for HIV prevention. AIDS Patient Care STDS. 2012 Jul;26(7):395-405. doi: 10.1089/apc.2012.0030. Epub 2012 Jun 13. PMID 22694239
- [Background] Tripathi A, Ogbuanu C, Monger M, Gibson JJ, Duffus WA. Preexposure prophylaxis for HIV infection: healthcare providers' knowledge, perception, and willingness to adopt future implementation in the southern US. South Med J. 2012 Apr;105(4):199-206. doi: 10.1097/SMJ.0b013e31824f1a1b. PMID 22475669
- [Background] Guidance on Pre-Exposure Oral Prophylaxis (PrEP) for Serodiscordant Couples, Men and Transgender Women Who Have Sex with Men at High Risk of HIV: Recommendations for Use in the Context of Demonstration Projects. Geneva: World Health Organization; 2012 Jul. Available from http://www.ncbi.nlm.nih.gov/books/NBK132003/ PMID 23586123
- [Background] Beyrer C, Bekker LG, Pozniak A, Barre-Sinoussi F. Pre-exposure prophylaxis works--it's time to deliver. Lancet. 2015 Apr 18;385(9977):1482-4. doi: 10.1016/S0140-6736(15)60724-3. No abstract available. PMID 25933264
- [Background] Kirby T, Thornber-Dunwell M. Uptake of PrEP for HIV slow among MSM. Lancet. 2014 Feb 1;383(9915):399-400. doi: 10.1016/s0140-6736(14)60137-9. No abstract available. PMID 24494225
- [Background] Flash C, Landovitz R, Giler RM, Ng L, Magnuson D, Wooley SB, Rawlings K. Two years of Truvada for pre-exposure prophylaxis utilization in the US. J Int AIDS Soc. 2014 Nov 2;17(4 Suppl 3):19730. doi: 10.7448/IAS.17.4.19730. eCollection 2014. PMID 25397476
- [Background] Liu A, Cohen S, Follansbee S, Cohan D, Weber S, Sachdev D, Buchbinder S. Early experiences implementing pre-exposure prophylaxis (PrEP) for HIV prevention in San Francisco. PLoS Med. 2014 Mar 4;11(3):e1001613. doi: 10.1371/journal.pmed.1001613. eCollection 2014 Mar. PMID 24595035
- [Background] King HL, Keller SB, Giancola MA, Rodriguez DA, Chau JJ, Young JA, Little SJ, Smith DM. Pre-exposure prophylaxis accessibility research and evaluation (PrEPARE Study). AIDS Behav. 2014 Sep;18(9):1722-5. doi: 10.1007/s10461-014-0845-5. PMID 25017425
- [Background] Cohen SE, Vittinghoff E, Bacon O, Doblecki-Lewis S, Postle BS, Feaster DJ, Matheson T, Trainor N, Blue RW, Estrada Y, Coleman ME, Elion R, Castro JG, Chege W, Philip SS, Buchbinder S, Kolber MA, Liu AY. High interest in preexposure prophylaxis among men who have sex with men at risk for HIV infection: baseline data from the US PrEP demonstration project. J Acquir Immune Defic Syndr. 2015 Apr 1;68(4):439-48. doi: 10.1097/QAI.0000000000000479. PMID 25501614
- [Background] McDougal SJ, Alexander J, Dhanireddy S, Harrington RD, Stekler JD. Non-occupational post-exposure prophylaxis for HIV: 10-year retrospective analysis in Seattle, Washington. PLoS One. 2014 Aug 20;9(8):e105030. doi: 10.1371/journal.pone.0105030. eCollection 2014. PMID 25140868
- [Background] Centers for Disease Control and Prevention (CDC). Interim guidance: preexposure prophylaxis for the prevention of HIV infection in men who have sex with men. MMWR Morb Mortal Wkly Rep. 2011 Jan 28;60(3):65-8. PMID 21270743
- [Background] Norton WE, Larson RS, Dearing JW. Primary care and public health partnerships for implementing pre-exposure prophylaxis. Am J Prev Med. 2013 Jan;44(1 Suppl 2):S77-9. doi: 10.1016/j.amepre.2012.09.037. No abstract available. PMID 23253766
- [Background] Castel AD, Feaster DJ, Tang W, Willis S, Jordan H, Villamizar K, Kharfen M, Kolber MA, Rodriguez A, Metsch LR. Understanding HIV Care Provider Attitudes Regarding Intentions to Prescribe PrEP. J Acquir Immune Defic Syndr. 2015 Dec 15;70(5):520-8. doi: 10.1097/QAI.0000000000000780. PMID 26247895
- [Background] Morin SF, Yamey G, Rutherford GW. HIV pre-exposure prophylaxis. BMJ. 2012 Aug 13;345:e5412. doi: 10.1136/bmj.e5412. No abstract available. PMID 22890030
- [Background] Campbell JD, Herbst JH, Koppenhaver RT, Smith DK. Antiretroviral prophylaxis for sexual and injection drug use acquisition of HIV. Am J Prev Med. 2013 Jan;44(1 Suppl 2):S63-9. doi: 10.1016/j.amepre.2012.09.045. PMID 23253764
- [Background] Grant RM, Anderson PL, McMahan V, Liu A, Amico KR, Mehrotra M, Hosek S, Mosquera C, Casapia M, Montoya O, Buchbinder S, Veloso VG, Mayer K, Chariyalertsak S, Bekker LG, Kallas EG, Schechter M, Guanira J, Bushman L, Burns DN, Rooney JF, Glidden DV; iPrEx study team. Uptake of pre-exposure prophylaxis, sexual practices, and HIV incidence in men and transgender women who have sex with men: a cohort study. Lancet Infect Dis. 2014 Sep;14(9):820-9. doi: 10.1016/S1473-3099(14)70847-3. Epub 2014 Jul 22. PMID 25065857
- [Background] Baeten JM, Donnell D, Ndase P, Mugo NR, Campbell JD, Wangisi J, Tappero JW, Bukusi EA, Cohen CR, Katabira E, Ronald A, Tumwesigye E, Were E, Fife KH, Kiarie J, Farquhar C, John-Stewart G, Kakia A, Odoyo J, Mucunguzi A, Nakku-Joloba E, Twesigye R, Ngure K, Apaka C, Tamooh H, Gabona F, Mujugira A, Panteleeff D, Thomas KK, Kidoguchi L, Krows M, Revall J, Morrison S, Haugen H, Emmanuel-Ogier M, Ondrejcek L, Coombs RW, Frenkel L, Hendrix C, Bumpus NN, Bangsberg D, Haberer JE, Stevens WS, Lingappa JR, Celum C; Partners PrEP Study Team. Antiretroviral prophylaxis for HIV prevention in heterosexual men and women. N Engl J Med. 2012 Aug 2;367(5):399-410. doi: 10.1056/NEJMoa1108524. Epub 2012 Jul 11. PMID 22784037
- [Background] Molina JM, Pintado C, Gatey C, Ponscarme D, Charbonneau P, Loze B, Rozenbaum W, Delaugerre C. Challenges and opportunities for oral pre-exposure prophylaxis in the prevention of HIV infection: where are we in Europe? BMC Med. 2013 Aug 23;11:186. doi: 10.1186/1741-7015-11-186. PMID 23972284
- [Background] Hosek SG, Siberry G, Bell M, Lally M, Kapogiannis B, Green K, Fernandez MI, Rutledge B, Martinez J, Garofalo R, Wilson CM; Adolescent Trials Network for HIVAIDS Interventions (ATN). The acceptability and feasibility of an HIV preexposure prophylaxis (PrEP) trial with young men who have sex with men. J Acquir Immune Defic Syndr. 2013 Apr 1;62(4):447-56. doi: 10.1097/QAI.0b013e3182801081. PMID 24135734
- [Background] Mayer KH, Krakower DS. Editorial Commentary: Scaling Up Antiretroviral Preexposure Prophylaxis: Moving From Trials to Implementation. Clin Infect Dis. 2015 Nov 15;61(10):1598-600. doi: 10.1093/cid/civ665. Epub 2015 Aug 13. No abstract available. PMID 26270688
- [Background] Kelley CF, Kahle E, Siegler A, Sanchez T, Del Rio C, Sullivan PS, Rosenberg ES. Applying a PrEP Continuum of Care for Men Who Have Sex With Men in Atlanta, Georgia. Clin Infect Dis. 2015 Nov 15;61(10):1590-7. doi: 10.1093/cid/civ664. Epub 2015 Aug 13. PMID 26270691
- [Background] Brooks RA, Landovitz RJ, Regan R, Lee SJ, Allen VC Jr. Perceptions of and intentions to adopt HIV pre-exposure prophylaxis among black men who have sex with men in Los Angeles. Int J STD AIDS. 2015 Dec;26(14):1040-8. doi: 10.1177/0956462415570159. Epub 2015 Jan 30. PMID 25638214
- [Background] Eaton LA, Driffin DD, Bauermeister J, Smith H, Conway-Washington C. Minimal Awareness and Stalled Uptake of Pre-Exposure Prophylaxis (PrEP) Among at Risk, HIV-Negative, Black Men Who Have Sex with Men. AIDS Patient Care STDS. 2015 Aug;29(8):423-9. doi: 10.1089/apc.2014.0303. Epub 2015 Jun 17. PMID 26083143
- [Background] Thorpe KE, Zwarenstein M, Oxman AD, Treweek S, Furberg CD, Altman DG, Tunis S, Bergel E, Harvey I, Magid DJ, Chalkidou K. A pragmatic-explanatory continuum indicator summary (PRECIS): a tool to help trial designers. CMAJ. 2009 May 12;180(10):E47-57. doi: 10.1503/cmaj.090523. Epub 2009 Apr 16. No abstract available. PMID 19372436
- [Background] Bauman LJ, Braunstein S, Calderon Y, Chhabra R, Cutler B, Leider J, Rivera A, Sclafane J, Tsoi B, Watnick D. Barriers and facilitators of linkage to HIV primary care in New York City. J Acquir Immune Defic Syndr. 2013 Nov 1;64 Suppl 1(0 1):S20-6. doi: 10.1097/QAI.0b013e3182a99c19. PMID 24126445
- [Background] Remien RH, Bauman LJ, Mantell JE, Tsoi B, Lopez-Rios J, Chhabra R, DiCarlo A, Watnick D, Rivera A, Teitelman N, Cutler B, Warne P. Barriers and facilitators to engagement of vulnerable populations in HIV primary care in New York City. J Acquir Immune Defic Syndr. 2015 May 1;69 Suppl 1(0 1):S16-24. doi: 10.1097/QAI.0000000000000577. PMID 25867774
- [Background] Diiorio CA, Kobau R, Holden EW, Berkowitz JM, Kamin SL, Antonak RF, Austin JK, Baker GA, Bauman LJ, Gilliam F, Thurman DJ, Price PH. Developing a measure to assess attitudes toward epilepsy in the US population. Epilepsy Behav. 2004 Dec;5(6):965-75. doi: 10.1016/j.yebeh.2004.08.020. PMID 15582846
- [Background] Crain EF, Mortimer KM, Bauman LJ, Kercsmar CM, Weiss KB, Wissow L, Mitchell H, Rotor D. Pediatric asthma care in the emergency department: measuring the quality of history-taking and discharge planning. J Asthma. 1999;36(1):129-38. doi: 10.3109/02770909909065156. PMID 10077142
- [Background] Okun A, Stein RE, Bauman LJ, Silver EJ. Content validity of the Psychiatric Symptom Index, CES-depression Scale, and State-Trait Anxiety Inventory from the perspective of DSM-IV. Psychol Rep. 1996 Dec;79(3 Pt 1):1059-69. doi: 10.2466/pr0.1996.79.3.1059. PMID 8969117
- [Background] Pequegnat W, Szacpocznik J, Bauman LJ, et al. Measurement relevant to the role of families in prevention and adaptation to HIV/AIDS. AIDS and Behavior. 2001;5(1):1-19.
- [Background] Bauman LJ, Wright E, Leickly FE, Crain E, Kruszon-Moran D, Wade SL, Visness CM. Relationship of adherence to pediatric asthma morbidity among inner-city children. Pediatrics. 2002 Jul;110(1 Pt 1):e6. doi: 10.1542/peds.110.1.e6. PMID 12093987
- [Background] Stein RE, Westbrook LE, Bauman LJ. The Questionnaire for Identifying Children with Chronic Conditions: a measure based on a noncategorical approach. Pediatrics. 1997 Apr;99(4):513-21. doi: 10.1542/peds.99.4.513. PMID 9093290
- [Background] Stein RE, Bauman LJ, Epstein SG, Gardner JD, Walker DK. How well does the questionnaire for identifying children with chronic conditions identify individual children who have chronic conditions? Arch Pediatr Adolesc Med. 2000 May;154(5):447-52. doi: 10.1001/archpedi.154.5.447. PMID 10807293
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Bronfenbrenner U, Ceci SJ. Nature-nurture reconceptualized in developmental perspective: a bioecological model. Psychol Rev. 1994 Oct;101(4):568-86. doi: 10.1037/0033-295x.101.4.568. PMID 7984707
- [Background] Ajzen I, The theory of planned behavior. Organizational Behavior and Human Decision Process. 1991;50(2):179-211
- [Background] Ajzen I, Madden TJ. Prediction of goal-directed behavior: attitudes, intentions, and perceived behavioral control. Journal of Experimental Social Psychology. 1986;22(5):453-474
- [Background] Bandura A. Human agency in social cognitive theory. Am Psychol. 1989 Sep;44(9):1175-84. doi: 10.1037/0003-066x.44.9.1175. PMID 2782727
- [Background] Greenhalgh T, Robert G, Macfarlane F, Bate P, Kyriakidou O. Diffusion of innovations in service organizations: systematic review and recommendations. Milbank Q. 2004;82(4):581-629. doi: 10.1111/j.0887-378X.2004.00325.x. PMID 15595944
- [Background] Carlfjord S, Lindberg M, Bendtsen P, Nilsen P, Andersson A. Key factors influencing adoption of an innovation in primary health care: a qualitative study based on implementation theory. BMC Fam Pract. 2010 Aug 23;11:60. doi: 10.1186/1471-2296-11-60. PMID 20731817
- [Background] Davis D, O'Brien MA, Freemantle N, Wolf FM, Mazmanian P, Taylor-Vaisey A. Impact of formal continuing medical education: do conferences, workshops, rounds, and other traditional continuing education activities change physician behavior or health care outcomes? JAMA. 1999 Sep 1;282(9):867-74. doi: 10.1001/jama.282.9.867. PMID 10478694
- [Background] Drainoni ML, Dekker D, Lee-Hood E, Boehmer U, Relf M. HIV medical care provider practices for reducing high-risk sexual behavior: results of a qualitative study. AIDS Patient Care STDS. 2009 May;23(5):347-56. doi: 10.1089/apc.2008.0063. PMID 19413497
- [Background] Morin SF, Koester KA, Steward WT, Maiorana A, McLaughlin M, Myers JJ, Vernon K, Chesney MA. Missed opportunities: prevention with HIV-infected patients in clinical care settings. J Acquir Immune Defic Syndr. 2004 Aug 1;36(4):960-6. doi: 10.1097/00126334-200408010-00010. PMID 15220703
- [Background] Epstein RM, Morse DS, Frankel RM, Frarey L, Anderson K, Beckman HB. Awkward moments in patient-physician communication about HIV risk. Ann Intern Med. 1998 Mar 15;128(6):435-42. doi: 10.7326/0003-4819-128-6-199803150-00003. PMID 9499326
- [Background] Mimiaga MJ, Goldhammer H, Belanoff C, Tetu AM, Mayer KH. Men who have sex with men: perceptions about sexual risk, HIV and sexually transmitted disease testing, and provider communication. Sex Transm Dis. 2007 Feb;34(2):113-9. doi: 10.1097/01.olq.0000225327.13214.bf. PMID 16810121
- [Background] Flodgren G, Parmelli E, Doumit G, Gattellari M, O'Brien MA, Grimshaw J, Eccles MP. Local opinion leaders: effects on professional practice and health care outcomes. Cochrane Database Syst Rev. 2011 Aug 10;(8):CD000125. doi: 10.1002/14651858.CD000125.pub4. PMID 21833939
- [Background] Nair H, Manchanda P, Bhatia T. Asymmetric social interactions in physician prescription behavior: The role of opinion Leaders. Journal of Marketing Research 47(5): 883-895, 2010.
- [Background] Majumdar SR, Tsuyuki RT, McAlister FA. Impact of opinion leader-endorsed evidence summaries on the quality of prescribing for patients with cardiovascular disease: a randomized controlled trial. Am Heart J. 2007 Jan;153(1):22.e1-8. doi: 10.1016/j.ahj.2006.07.030. PMID 17174632
- [Background] Hettema J, Steele J, Miller WR. Motivational interviewing. Annu Rev Clin Psychol. 2005;1:91-111. doi: 10.1146/annurev.clinpsy.1.102803.143833. PMID 17716083
- [Background] Exner TM, Mantell JE, Adeokun LA, Udoh IA, Ladipo OA, Delano GE, Faleye J, Akinpelu K. Mobilizing men as partners: the results of an intervention to increase dual protection among Nigerian men. Health Educ Res. 2009 Oct;24(5):846-54. doi: 10.1093/her/cyp021. Epub 2009 Apr 9. PMID 19359352
- [Background] Mantell JE, Exner TM, Cooper D, Bai D, Leu CS, Hoffman S, Myer L, Moodley J, Kelvin EA, Constant D, Jennings K, Zweigenthal V, Stein ZA. Pregnancy intent among a sample of recently diagnosed HIV-positive women and men practicing unprotected sex in Cape Town, South Africa. J Acquir Immune Defic Syndr. 2014 Dec 1;67 Suppl 4(Suppl 4):S202-9. doi: 10.1097/QAI.0000000000000369. PMID 25436819
- [Background] Smith DK, Pals SL, Herbst JH, Shinde S, Carey JW. Development of a clinical screening index predictive of incident HIV infection among men who have sex with men in the United States. J Acquir Immune Defic Syndr. 2012 Aug 1;60(4):421-7. doi: 10.1097/QAI.0b013e318256b2f6. PMID 22487585
- [Background] Flynn NM, Forthal DN, Harro CD, Judson FN, Mayer KH, Para MF; rgp120 HIV Vaccine Study Group. Placebo-controlled phase 3 trial of a recombinant glycoprotein 120 vaccine to prevent HIV-1 infection. J Infect Dis. 2005 Mar 1;191(5):654-65. doi: 10.1086/428404. Epub 2005 Jan 27. PMID 15688278
- [Background] Bartholow BN, Buchbinder S, Celum C, Goli V, Koblin B, Para M, Marmor M, Novak RM, Mayer K, Creticos C, Orozco-Cronin P, Popovic V, Mastro TD; VISION/VAX004 Study Team. HIV sexual risk behavior over 36 months of follow-up in the world's first HIV vaccine efficacy trial. J Acquir Immune Defic Syndr. 2005 May 1;39(1):90-101. doi: 10.1097/01.qai.0000143600.41363.78. PMID 15851919
- [Background] Koblin B, Chesney M, Coates T; EXPLORE Study Team. Effects of a behavioural intervention to reduce acquisition of HIV infection among men who have sex with men: the EXPLORE randomised controlled study. Lancet. 2004 Jul 3-9;364(9428):41-50. doi: 10.1016/S0140-6736(04)16588-4. PMID 15234855
- [Background] Celum C, Baeten JM. Tenofovir-based pre-exposure prophylaxis for HIV prevention: evolving evidence. Curr Opin Infect Dis. 2012 Feb;25(1):51-7. doi: 10.1097/QCO.0b013e32834ef5ef. PMID 22156901
- [Background] Kahle EM, Hughes JP, Lingappa JR, John-Stewart G, Celum C, Nakku-Joloba E, Njuguna S, Mugo N, Bukusi E, Manongi R, Baeten JM; Partners in Prevention HSVHIV Transmission Study and the Partners PrEP Study Teams. An empiric risk scoring tool for identifying high-risk heterosexual HIV-1-serodiscordant couples for targeted HIV-1 prevention. J Acquir Immune Defic Syndr. 2013 Mar 1;62(3):339-47. doi: 10.1097/QAI.0b013e31827e622d. PMID 23187945
- [Background] Nadeem E, Olin SS, Hill LC, Hoagwood KE, Horwitz SM. Understanding the components of quality improvement collaboratives: a systematic literature review. Milbank Q. 2013 Jun;91(2):354-94. doi: 10.1111/milq.12016. PMID 23758514
- [Background] Palesch YY, Tilley BC. An efficient multi-stage, single-arm Phase II futility design for ALS. Amyotroph Lateral Scler Other Motor Neuron Disord. 2004 Sep;5 Suppl 1:55-6. doi: 10.1080/17434470410020003. No abstract available. PMID 15512874
- [Background] Levin B. The utility of futility. Stroke. 2005 Nov;36(11):2331-2. doi: 10.1161/01.STR.0000185722.99167.56. Epub 2005 Oct 13. No abstract available. PMID 16224096
- [Background] Collins LM, Murphy SA, Strecher V. The multiphase optimization strategy (MOST) and the sequential multiple assignment randomized trial (SMART): new methods for more potent eHealth interventions. Am J Prev Med. 2007 May;32(5 Suppl):S112-8. doi: 10.1016/j.amepre.2007.01.022. PMID 17466815
- [Background] Cook PF, Friedman R, Lord A, Bradley-Springer LA. Outcomes of multimodal training for healthcare professionals at an AIDS education and training center. Eval Health Prof. 2009 Mar;32(1):3-22. doi: 10.1177/0163278708328736. Epub 2009 Jan 8. PMID 19131377
- [Background] Kelly JA, Somlai AM, DiFranceisco WJ, Otto-Salaj LL, McAuliffe TL, Hackl KL, Heckman TG, Holtgrave DR, Rompa D. Bridging the gap between the science and service of HIV prevention: transferring effective research-based HIV prevention interventions to community AIDS service providers. Am J Public Health. 2000 Jul;90(7):1082-8. doi: 10.2105/ajph.90.7.1082. PMID 10897186
- [Background] Kelly JA, Somlai AM, Benotsch EG, McAuliffe TL, Amirkhanian YA, Brown KD, Stevenson LY, Fernandez MI, Sitzler C, Gore-Felton C, Pinkerton SD, Weinhardt LS, Opgenorth KM. Distance communication transfer of HIV prevention interventions to service providers. Science. 2004 Sep 24;305(5692):1953-5. doi: 10.1126/science.1100733. PMID 15448268
- [Background] Wilson IB, Fowler FJ Jr, Cosenza CA, Michaud J, Bentkover J, Rana A, Kogelman L, Rogers WH. Cognitive and field testing of a new set of medication adherence self-report items for HIV care. AIDS Behav. 2014 Dec;18(12):2349-58. doi: 10.1007/s10461-013-0610-1. PMID 24077970
- [Background] Vanable PA, Ostrow DG, McKirnan DJ. Viral load and HIV treatment attitudes as correlates of sexual risk behavior among HIV-positive gay men. J Psychosom Res. 2003 Mar;54(3):263-9. doi: 10.1016/s0022-3999(02)00483-x. PMID 12614836
- [Background] Castillo-Mancilla JR, Zheng JH, Rower JE, Meditz A, Gardner EM, Predhomme J, Fernandez C, Langness J, Kiser JJ, Bushman LR, Anderson PL. Tenofovir, emtricitabine, and tenofovir diphosphate in dried blood spots for determining recent and cumulative drug exposure. AIDS Res Hum Retroviruses. 2013 Feb;29(2):384-90. doi: 10.1089/AID.2012.0089. Epub 2012 Oct 10. PMID 22935078
- [Background] Karasz A, Singelis TM. Qualitative and Mixed Methods Research in Cross-cultural Psychology: Introduction to the Special Issue. J Cross Cult Psychol. 2009 Nov 1;40(6):909-916. doi: 10.1177/0022022109349172. No abstract available. PMID 21666752
- [Background] Hollway W, Jefferson T. Eliciting narrative through the in-depth interview. Qualitative Inquiry. 3(1): 53-70, 1997.
- [Background] Ware NC, Wyatt MA, Haberer JE, Baeten JM, Kintu A, Psaros C, Safren S, Tumwesigye E, Celum CL, Bangsberg DR. What's love got to do with it? Explaining adherence to oral antiretroviral pre-exposure prophylaxis for HIV-serodiscordant couples. J Acquir Immune Defic Syndr. 2012 Apr 15;59(5):463-8. doi: 10.1097/QAI.0b013e31824a060b. PMID 22267018
- [Background] Corneli AL, McKenna K, Perry B, Ahmed K, Agot K, Malamatsho F, Skhosana J, Odhiambo J, Van Damme L. The science of being a study participant: FEM-PrEP participants' explanations for overreporting adherence to the study pills and for the whereabouts of unused pills. J Acquir Immune Defic Syndr. 2015 Apr 15;68(5):578-84. doi: 10.1097/QAI.0000000000000525. PMID 25761233
- [Background] Mimiaga MJ, White JM, Krakower DS, Biello KB, Mayer KH. Suboptimal awareness and comprehension of published preexposure prophylaxis efficacy results among physicians in Massachusetts. AIDS Care. 2014;26(6):684-93. doi: 10.1080/09540121.2013.845289. Epub 2013 Oct 14. PMID 24116985
- [Background] Tellalian D, Maznavi K, Bredeek UF, Hardy WD. Pre-exposure prophylaxis (PrEP) for HIV infection: results of a survey of HIV healthcare providers evaluating their knowledge, attitudes, and prescribing practices. AIDS Patient Care STDS. 2013 Oct;27(10):553-9. doi: 10.1089/apc.2013.0173. Epub 2013 Sep 20. PMID 24053478
- [Background] Karris MY, Beekmann SE, Mehta SR, Anderson CM, Polgreen PM. Are we prepped for preexposure prophylaxis (PrEP)? Provider opinions on the real-world use of PrEP in the United States and Canada. Clin Infect Dis. 2014 Mar;58(5):704-12. doi: 10.1093/cid/cit796. Epub 2013 Dec 6. PMID 24319083
- See also: Office of National AIDS Policy. The White House. National HIV/AIDS Strategy for the United States — https://obamawhitehouse.archives.gov/sites/default/files/uploads/NHAS.pdf
- See also: Office of National AIDS Policy. The White House. National HIV/AIDS Strategy: Implementation Update — https://obamawhitehouse.archives.gov/sites/default/files/uploads/hiv_aids_july_2011.pdf
- See also: NIH HIV/AIDS Research Priorities and Guidelines for Determining AIDS Funding — https://grants.nih.gov/grants/guide/notice-files/NOT-OD-15-137.html
- See also: Mera R, Rawlings M, Pechonkina A, et al. Status of Truvada (TVD) for HIV Pre-Exposure Prophylaxis (PrEP) in the United States: An Early Drug Utilization Analysis — http://www.natap.org/2013/ICAAC/ICAAC_18.htm
- See also: Glidden D, Buchbinder S, Anderson P, et al. PrEP Engagement for HIV Prevention: Results From the iPrEx Open Label Extension (OLE) — http://www.croiconference.org/sessions/prep-engagement-hiv-prevention-results-iprex-open-label-extension-ole
- See also: McCormack S, Dunn D. Pragmatic Open-Label Randomised Trial of Preexposure Prophylaxis: The PROUD Study — http://www.croiconference.org/sessions/pragmatic-open-label-randomised-trial-preexposure-prophylaxis-proud-study
- See also: Molina J-M, Capitant C, Spire B, et al. On Demand PrEP With Oral TDF-FTC in MSM: Results of the ANRS Ipergay Trial — http://www.croiconference.org/sessions/demand-prep-oral-tdf-ftc-msm-results-anrs-ipergay-trial
- See also: Agency for Quality Healthcare Research and Quality. Translating Research Into Practice (TRIP)-II — https://archive.ahrq.gov/research/findings/factsheets/translating/tripfac/trip2fac.html
- See also: Strategies for Using Pre-Exposure Prophylaxis (PrEP) to Lower HIV Incidence in Select Populations — http://www.theaidsinstitute.org/sites/default/files/attachments/PrEP%20implementation%20strategies%20document.pdf
- See also: Murcury News, June 2012. FDA delays decision on Gilead drug that could prevent HIV. — https://www.mercurynews.com/2012/06/08/fda-delays-decision-on-gilead-drug-that-could-prevent-hiv/
- See also: Solutions PH. HIV prevention programs: RFA issued by Public Health Solutions on behalf lf the New York City Department of Health and Mental Hygiene. Bureau of HIV/AIDS Prevention and Control. March 15, 2015 — http://www.healthsolutions.org
- See also: New York City Department of Health and Mental Hygiene. New York City HIV/AIDS Annual Surveillance Statistics 2011 — https://www1.nyc.gov/assets/doh/downloads/pdf/ah/surveillance2011-table-all.pdf
- See also: New York City Department of Health and Mental Hygiene. Epiquery: New York City Interactive Health Data System - New York City Community Health Survey 2011 [HIV testing, condom use frequency (anal sex)]. — https://a816-healthpsi.nyc.gov/epiquery/CHS/CHSXIndex.html
- See also: New York City Department of Health and Human Hygiene. NYC HIV/AIDS Surveillance Statistics — https://www1.nyc.gov/site/doh/data/data-sets/hiv-aids-annual-surveillance-statistics.page
- See also: Health Resource and Service Administration. Primary Care: The Health Center Program 2012 — https://bphc.hrsa.gov/programrequirements/index.html
- See also: HealthKeep — http://www.healthkeep.com
- See also: Crunch T. HealthKeep launches an anonymous social network to let you share and track health information. April 16, 2013. — https://techcrunch.com/2013/04/16/healthkeep-launches-an-anonymous-social-network-to-let-you-share-and-track-health-information/
- See also: Sense Health — https://sensehealth.com
- See also: Randomized Control Trial Finds Sense Health's Mobile Care Management Platform Can Boost Patient Adherence. July 9, 2014 — https://www.prnewswire.com/news-releases/randomized-control-trial-finds-sense-healths-mobile-care-management-platform-can-boost-patient-adherence-266414041.html
- See also: Dedoose. Dedoose Qualitative Software. Sociocultural Research Consultants, LLC. 2011. — https://www.dedoose.com/